CLINICAL TRIAL: NCT03420274
Title: Ensuring Patients' Informed Access to Noninvasive Prenatal Testing
Acronym: NEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Indiana University (Other); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-987; R01HG010092 (NIH)
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Genetic Disease; Genetic Syndrome; Prenatal Disorder; Prenatal Maternal Abnormality; Pregnancy Complications
Keywords: Shared decision-making; Prenatal genetic testing; Noninvasive prenatal testing (NIPT); Cell free fetal DNA (cfDNA); Informed consent
MeSH Terms: conditions — Genetic Diseases, Inborn; Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: This will be a cluster randomized trial examining a shared decision-making intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will utilize a point-of-care shared decision-making tool (NEST).
  Interventions: Behavioral: NEST
- Control (Placebo Comparator): This group will utilize usual care with respect to healthcare provider practice for education and counseling.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: NEST — This is a point-of-care shared decision-making instrument.
  Arms: Intervention
Behavioral: Usual care — This group will utilize usual care with respect to healthcare provider practice for education and counseling.
  Arms: Control

SUMMARY:
Noninvasive prenatal genetic testing (NIPT) is an important new screening test option provided to pregnant women in the first trimester of pregnancy. The advantage of this screen is that is provides information about the risk of trisomy 13, trisomy 18, and trisomy 21 with greater accuracy than conventional screens. At the same time, NIPT can produce information about the risk of a cohort of other fetal genetic variants, including sex chromosome aneuploidies and microdeletion syndromes. While not yet clinically available for whole exome sequencing, the potential for this next clinical application already exists. The challenge is that, while this is an important new test, there are little data about how to best structure patient-centered decisions about its use, including decisions if to use this screen and how the information may directly inform subsequent prenatal care decisions. The purpose of this study is to gain formative data about current practice patterns with respect to how NIPT is discussed in the clinical visit and to use these data to help inform best practices for its continued use in the clinical setting.

DETAILED DESCRIPTION:
Noninvasive prenatal genetic testing (NIPT), also known as cell-free fetal DNA screening, has dramatically altered the delivery of prenatal care. Prior to NIPT, fetal aneuploidy risk was assessed using conventional screens, most commonly maternal serum screens (MSS, e.g. the Quadruple screen). While MSS provided information about the risk of trisomy (T) 21, T13, and T18, its use led to many false positive results which required amniocentesis or chorionic villus sampling to clarify. The risk of iatrogenic miscarriage from these diagnostic procedures is low, but the possibility of this consequence is a major driver in how healthcare providers and patients think about prenatal genetic risk and assessment. NIPT has significantly changed this long-standing paradigm. While not diagnostic, NIPT offers increased accuracy with lower false positive and false negative rates than MSS when screening for common autosomal aneuploidies. Unlike conventional screens, NIPT provides information never before a part of routine screening, such as the presence of sex chromosome aneuploidies (SCAs), microdeletions, and fetal sex. Already the capability exists to utilize NIPT in conjunction with whole exome sequencing to detect an unlimited number of fetal genomic variants, many with undetermined significance. The list of conditions that NIPT can screen for is expanding rapidly and has outpaced the rate at which evidence-based strategies for its integration can be developed and implemented.

Expectant parents must be prepared to make informed decisions about NIPT, including whether to use it and how to address the prenatal care decisions that result from that choice. For some, information from NIPT may inform the decision to undergo additional tests and either prepare for the birth of a child with a serious, potentially life-threatening condition, or end the pregnancy if a condition is confirmed by diagnostic testing. While this has been the case for all forms of prenatal testing, NIPT presents unique challenges to this decision-making process because it provides information about a series of conditions with variable phenotypic severity of which patients have little familiarity (e.g., Turner syndrome, Klinefelter syndrome), as well as providing information about markers of undetermined significance. As with conventional screening, there is the potential for a false positive or false negative result for each of these findings. Furthermore, information gained from NIPT may have unintended consequences by identifying maternal or paternal factors that may be unwanted or unexpected. Previous studies have demonstrated that expectant parents already face a number of challenges in obtaining accurate, unbiased in-formation and decisional support when navigating conventional prenatal genetic screens and diagnostic tests (abbreviated as "prenatal testing" in the rest of this document) and the consequences of being un-prepared for a positive test result. This situation has been exacerbated with the introduction of NIPT and will worsen with its expansion. Initially, NIPT was indicated for a subset of the obstetric population, namely women considered high-risk for aneuploidy due to advanced maternal age or reproductive history. Now, NIPT is becoming available for use by the general obstetric population as a primary screen. Clinicians will have to provide individualized counseling to pregnant patients about the advantages and dis-advantages of NIPT compared to other prenatal testing options. As part of this process, they will need to assist patients in placing this information in the context of their goals, values, and beliefs about parenthood, disability, and termination. The magnitude of the resulting challenge becomes evident when considering that over four million women receive prenatal care in the U.S. annually10 and there are not enough prenatal genetic counselors (GC) or maternal-fetal medicine specialists (MFM) to meet this demand, particularly in rural and urban settings that already face poorer obstetric outcomes due to barriers in access to prenatal care. It is unclear how the medical profession will respond to this unprecedented challenge.

The current situation places a heavy burden on primary obstetric (OB) providers to play a greater role in introducing patients to the option of NIPT and to facilitate decision-making about its use. Already, there are growing numbers of OB providers ordering NIPT, either with or without the involvement of a GC or a MFM, a trend that is expected to continue with the ongoing expansion of NIPT.39 Thus, an urgent clinical problem has emerged: there is a lack of evidence-based tools to guide OB providers in effective and individualized education and decision support for NIPT. To date, the focus of interventions has been on the development of decision aids and other educational resources to independently educate patients and OB providers about prenatal genetic assessment. These tools may impart information and provide a degree of decision support; however, they do not address the dynamic interaction that leads to the exchange of such information during the clinical visit. Data accrued from our recent work indicate that these strategies do not provide sufficient support or guidance about how to structure effective shared decision-making (SDM) discussions between the patient and OB provider. Studies, including work from our cur-rent R21, demonstrate that important barriers exist for patients seeking the information and support needed to navigate their prenatal testing options and make informed, value-reflective decisions about NIPT. While many women are familiar with common autosomal aneuploidies such as T21, they have little knowledge of SCAs and significantly less knowledge of microdeletion syndromes. Patients are over-whelmed by the prospect of learning enough about each of the different conditions that NIPT can detect. As a result, women increasingly rely upon guidance from OB providers with whom they have an established relationship to help determine which, if any, prenatal testing option to utilize. These are important discussions that take place in the clinical encounter and which educational modules and decision aids alone cannot sufficiently replace. Barriers also exist for OB providers, who report uncertainty about how to provide personalized, effective, and patient-centered counseling about NIPT, particularly under conditions of limited time, reimbursement for counseling, and resources to meet the needs of a diverse population of patients with varying degrees of health literacy and knowledge of genetic conditions, as well as different beliefs about parenthood, disability, and pregnancy termination. Current educational and counseling efforts used by OB providers may not be meeting the self-reported educational needs and decision-making preferences of patients considering NIPT, particularly those pertaining to personal values. Moreover, both patients and providers are concerned about being negatively judged or stereo-typed in discussing topics related to pregnancy termination and infant/child disability, particularly as NIPT increasingly identifies conditions with a range of phenotypes.

The delivery of high-quality, evidence-based prenatal care and access to NIPT will only occur if patients have information and support to make informed, values-based choices about their prenatal testing options. Given the relationship of informed decision-making with healthcare quality, access, and outcomes, it is critical to have effective, evidence-based mechanisms that are responsive to the needs and priorities of patients, the day-to-day challenges faced by providers, and the current scientific evidence and clinical practice guidelines about NIPT. While it is recognized that providers should involve patients in healthcare by means of a SDM process, how to achieve that level of communication within the constraints and challenges of the practice of obstetrics remains unknown. Thus, the goal of this study is to conduct a cluster, randomized trial to test an evidence-based tool termed NEST (for NIPT Education Sup-port Tool) to support patients' decision-making, focusing on the communication that takes place in the clinical encounter. The investigators will also identify aspects of the patient-provider interaction that are key to implementing effective strategies responsive to the challenges posed by the continued development of NIPT. Our hypothesis is that, by focusing on the dynamic interaction between the patient and provider, NEST will result in a SDM process that, in turn, will both increase patients' ability to make an informed choice about NIPT and decrease the decisional conflict associated with that choice. The expected outcome of this study is a clinically relevant, point-of-care tool that can be utilized among a diverse group of patients and providers to facilitate decisions that are informed, consistent with the patient's values, and with which patients do not experience decisional conflict.

The investigators will recruit three groups: 1) pregnant women, 2) partners of pregnant women, and 3) prenatal healthcare providers. Randomization will occur at the level of the healthcare provider. Pregnant women will be randomized per their prenatal healthcare provider to NEST (intervention) or usual care (control).

The investigators anticipate that this study's findings will ultimately contribute to improving the quality of prenatal care by empowering pregnant women to make informed choices that reflect their needs and preferences as individuals and parents. The investigators also anticipate that OB providers will feel more prepared and confident when approaching conversations about NIPT.

ELIGIBILITY:
I. Pregnant women

Inclusion criteria:

1. 18 years of age or older
2. Present for their initial prenatal visit care with one of the providers enrolled in the study
3. Able to provide consent to participate in the study
4. Available for a follow up in the 1st or 2nd trimester of pregnancy
5. Have a viable intrauterine pregnancy
6. Present for care between 7-12 weeks estimated gestation age (EGA)

Since criteria 5 and 6 will not be determined until the conclusion of the first prenatal visit, women who meet criteria 1-4 will be eligible for participation.

Exclusion Criteria:

Women who are:

1. Less than 18 years of age
2. Not currently pregnant or an intrauterine pregnancy has not yet been established
3. Inability to provide informed consent for research participation

II. Self-identified partners of pregnant women

Inclusion criteria:

1. 18 years of age or older
2. The male or female partner (such as partner or mother/aunt/grandmother serving in the role of primary collaborative decision-maker in place of a partner) of a pregnant woman who has participated in the research
3. Participating in decision-making about the pregnancy
4. Ability to read and speak English
5. Ability to provide informed consent for research participation

Exclusion criteria:

1. Younger than 18 years of age
2. Not currently involved in the pregnancy or decision-making about prenatal care
3. Inability to speak or read English
4. Inability to provide informed consent for research participation

III. Prenatal healthcare providers

Inclusion criteria:

1. Board certified or board-eligible CNM, OB/GYNs or MFMs
2. Deliver outpatient prenatal care at one of the regional practices of the Cleveland Clinic
3. Able to read and speak English
4. Able to provide consent for research participation

Exclusion criteria:

1. OB/GYNs who do not currently provide prenatal care
2. Medical students, residents, and fellows
3. Hospitalists who do not provide outpatient obstetric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators will recruit 1) pregnant women, 2) self-identified partners of pregnant women (not limited to male partner), and 3) prenatal healthcare providers.
Enrollment: 644 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Shared decision-making (SDM) | 40 weeks estimated gestational age
  This will be measured using the OPTIONS scale, a validated scale developed to measure different components of a shared decision-making process in a clinical encounter as part of a direct observation approach.

SECONDARY OUTCOMES:
Informed choice | 40 weeks estimated gestational age
  This will be measured using the Multidimensional Measure of Choice (MMIC). The MMIC, a well-established and validated instrument, measures informed choice with respect to prenatal testing by assessing four factors: (1) patient knowledge, (2) attitudes, and (3) deliberation of alternatives, advantages, and disadvantages, of different testing options in the context of (4) decision about test utilization. It has subsequently been modified and validated to assess informed choice for NIPT.
Decisional regret: | 40 weeks estimated gestational age
  This will be measured using the validated Decisional Conflict Scale (DCS).

CONTACTS AND LOCATIONS:
Overall Officials: Ruth M Farrell, M.D., M.A., Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No